CLINICAL TRIAL: NCT06980675
Title: Clinical and Microbiological Study on Local Application of an Ozonated Olive Oil Gel in the Periodontal Pockets: a Randomized Double-blind Trial.
Brief Title: Ozonized Olive Oil in the Treatment of Periodontal Pockets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Massimo Petruzzi, Clinical Professor of Odontostomatology, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7493
Record Dates: First submitted 2024-05-25; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Pocket
Keywords: Ozonated Olive Oil; Periodontal Pocket; Periodontal Disease
MeSH Terms: conditions — Periodontal Pocket; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Double-blind Intervention Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozonized Olive Oil Intervention Group (Experimental): It has been administrated in the form of gel once a week for three weeks
  Interventions: Device: Activated Ozonized Olive Oil Gel
- Placebo Controlled Group (Placebo Comparator): Same description of Interventional Group
  Interventions: Other: Placebo gel

INTERVENTIONS:
Device: Activated Ozonized Olive Oil Gel — It is a natural oil which has been ozonized to improve the antimicrobial activity against periodontopathogenic bacterias
  Arms: Ozonized Olive Oil Intervention Group
Other: Placebo gel — Placebo gel with same texture, color, way of administration and taste of Activated Ozonized Olive Oil Gel
  Arms: Placebo Controlled Group

SUMMARY:
A randomized controlled clinical trial was conducted on 16 patients (8 males and 8 women) who were diagnosed chronic periodontitis. All the patients has been divided by randomization in two groups: control group treated with placebo gel and experimental group treated with gel based on ozonated EVO olive oil.

Both group after the evaluation of inclusion and exclusion criteria during the first visit, were subjected to hygiene treatment of removal tartar deposit, considered as standard of therapy for periodontitis.

After 15 days the hygiene treatment, patients were been randomized in two groups following the flow chart (t0) starting with: periodontal probing, microbiological samples and the first administration of gel. Next week (t1), has been collected the compliance and did the second administration of gel; the procedures will be the same also for another week (t2), until the last week (t3) when has been registered the second periodontal probing and did the second microbiological samples.

Data were collected to software Microsoft Excel and all the data analysis were conducted on this software to highlight significant differences between both groups. As the primary outcome was continuous variable and assuming normal distribution bilateral parametric test T-student was performed. An alpha error of 5% was considered, Beta error was not calculated as this was a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II, III, or IV periodontitis according to the new 2017 World Workshop periodontal classification
* Patients of either sex and older than 18 years of age
* Probing Pocket Depth (PPD) greater than or equal to 4 mm at 3 sites
* Patients who have signed consent to the study
* Collaborating patients

Exclusion Criteria:

* age < 18 years and/or inability to provide written informed consent;
* absence of family or social welfare support;
* non-drug-induced gingival hypertrophy,
* severe smokers (more than 20 cigarettes per day),
* consumers of high levels of alcohol,
* patients on corticosteroid treatment,
* diabetic patient,
* immunodepressive therapies,
* chemotherapies,
* radiotherapies,
* pregnancy states;
* lack of collaboration for ongoing postoperative reevaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Difference of Probing Pocket Depth (PPD) | One measure to assess inclusion, second mesure at randomization and third measure after 21 days
  It is a measures in mm assessed with periodontal probe in periodontal pockets

SECONDARY OUTCOMES:
Difference of Total microbial load | One measure at randomization and second measure after 21 days
  Expressed in percentage, samples performed with sterile paper cone and measurement performed with Applied Biosystem 7500 sequence detection system with Real Time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Petruzzi, PhD, MD, Principal Investigator — University of Bari
Locations (1):
- Odontostomatologic Departement of Policlinic of Bari, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT06980675/Prot_SAP_000.pdf